CLINICAL TRIAL: NCT05674292
Title: An Evaluation of the Effect of the Erchonia Corporation Violet Zerona® Z6 for Body Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-VZ6
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Circumference Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Erchonia Violet Zerona Z6 (Experimental): 405nm violet laser light therapy.
  Interventions: Device: Erchonia Violet Zerona Z6

INTERVENTIONS:
Device: Erchonia Violet Zerona Z6 — 405nm violet diode low level laser device

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® Violet Zerona Z6 (manufactured by Erchonia Corporation (the Company), an over-the-counter (OTC) laser device, in providing noninvasive body circumference reduction.

DETAILED DESCRIPTION:
The clinical study is an open-label non-inferiority design to evaluate the efficacy of the Erchonia® Violet Zerona Z6, an over-the-counter (OTC) laser device, in providing noninvasive circumference reduction. The clinical study protocol is based on the protocol for the clinical study whose results were submitted in support of clearance of the predicate device, the Erchonia® Zerona® Z6 OTC.

ELIGIBILITY:
Inclusion Criteria:

* BMI is 30 or less
* 18 years of age or older

Exclusion Criteria:

* Pregnant
* Open wounds (sores, cuts, ulcers, etc.)
* Individuals with or being treated for any cancerous growth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tracey Hishon, Bloomfield Hills, Michigan
  - Jamie Thayer, Marquette, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia Violet Zerona Z6
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia Violet Zerona Z6
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Combined Circumference Reduction in Inches of the Waist, Hips, and Bilateral Thighs
Description: Mean change in total combined circumference inches of the waist, hips and bilateral thighs from baseline to endpoint evaluation.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia Violet Zerona Z6
Number analyzed (Participants) | 25
inches | -3.91 (1.649)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Erchonia Violet Zerona Z6
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT05674292/Prot_SAP_ICF_000.pdf